CLINICAL TRIAL: NCT03239964
Title: Combined Surgical Excision and Intralesional Steroid Injection for Prevention of Post Caesarean Keloid Recurrence.A Randomized Controlled Trial.
Brief Title: Surgical Excision and Intralesional Steroid Injection for Prevention of Post Caesarean Keloid Recurrence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Amira S Dieb, Amira S Dieb, MD, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 88765510
Record Dates: First submitted 2017-07-29; First posted 2017-08-04 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Keloid
Keywords: recurrent keloid; surgical excision; steroids injection
MeSH Terms: conditions — Keloid | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- excision only group (Active Comparator): Under general or spinal anaesthesia done routinely during caesarean section, total extralesional surgical excision of keloid is performed and minimal undermining followed by usual steps of caesarean section. Primary closure of wound in layers is achieved in all cases. A running subcuticular prolene 2/0 stitch is used to suture the skin. Group A of 73 patients will not receive further injection. The wound is painted with betadine and sealed until postoperative day 14, at which time the subcuticular stitch is removed.
  Routine postoperative medications are given to all patients. They are advised to avoid direct sun exposure for the following month. No postoperative applications (eg, compression, steroid injections, etc) are used in any of the patients. All patients are reviewed once per month for 6 months.
  Interventions: Other: surgical excision
- excision and injection group (Active Comparator): Under general or spinal anaesthesia done routinely during caesarean section, total extralesional surgical excision of keloid is performed and minimal undermining followed by usual steps of caesarean section and primary closure of the wound in layers. A running subcuticular prolene 2/0 stitch is used to suture skin.In 73 patients (group B), wound edges are injected once with dexamethasone. A 1 mL syringe with a 30-gauge needle is used both intradermal and subdermal. Repeated alternate punctures are used to bathe the wound edges with the drug. Approximately 0.5-1 mL of dexamethasone (4 mg/mL) in wound tissue. The wound is painted with betadine and sealed until postoperative day 14 to remove the subcuticular stitch.
  Routine postoperative medications are given, avoidance of direct sun exposure for one month,No postoperative applications as compression, steroid injections, etc. All patients are reviewed once per month for 6 months.
  Interventions: Drug: Dexamethasone; Other: surgical excision

INTERVENTIONS:
Drug: Dexamethasone — the wound edges are injected once with dexamethasone. A 1 mL syringe with a 30-gauge needle is used and injection is both intradermal and subdermal. Repeated alternate punctures are used to bathe the wound edges with the drug. Approximately 0.5-1 mL of dexamethasone (4 mg/mL) in wound tissue.
  Arms: excision and injection group
Other: surgical excision — total extralesional surgical excision of the keloid is performed and minimal undermining

SUMMARY:
Two groups of patients (73 patients each) undergoing routine caesarean section has recurrent keloid at site of surgical scar. One group will undergo surgical excision of keloid. The other group will have combined surgical excision of keloid and single intralesional dexamethasone injection at edges of wound.All patients were reviewed once per month for 6 months for evidence of recurrence

DETAILED DESCRIPTION:
One hundred forty six patients that are admitted at Kasr Al Aini teaching university hospital for caesarean section, will be enrolled in this randomized clinical trial after approval by the local ethical health committee. A written informed consent will be obtained from each participant after full explanation of the procedure.

Under general or spinal anaesthesia done routinely during caesarean section, total extralesional surgical excision of the keloid is performed and minimal undermining followed by the usual steps of caesarean section. Primary closure of the wound in layers is achieved in all cases. A running subcuticular prolene 2/0 stitch is used to suture the skin. Group A of 73 patients will not receive further injection. In 73 patients (group B), the wound edges are injected once with dexamethasone. A 1 mL syringe with a 30-gauge needle is used and injection is both intradermal and subdermal. Repeated alternate punctures are used to bathe the wound edges with the drug. Approximately 0.5-1 mL of dexamethasone (4 mg/mL) in wound tissue.

For all patients, the wound is painted with betadine and sealed until postoperative day 14, at which time the subcuticular stitch is removed.

Postoperative medications are given to all patients in the form of analgesics and antibiotics as routinely given at the hospital. All patients were advised to avoid direct sun exposure for the following month. No postoperative applications (eg, compression, steroid injections, etc) were used in any of the patients. All patients were reviewed once per month for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented keloids of pfannenstiel incision or midline subumbilical incision of one to five years duration.
* Previous treatment of keloid and recurrence.
* Patient complaint of cosmetic disfiguring, pain or pruritis at site of scar.

Exclusion criteria:

* Scar <1 years' duration
* Scar extending beyond the limits of the original lesion
* postburn keloids
* Diabetes Mellitus, anaemia (haemoglobin level <10mg/dL), malignancy, malnutrition.
* local inflammation at site of scar
* Allergy to dexamethasone.
* Immunocompromized patients or patients on chronic steroid treatment.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with recurrent lesions | 6 months
  same/smaller/larger than pretreatment lesion

SECONDARY OUTCOMES:
Number of participantsc with pruritis | 6 months
  itching sensation at the site of wound
Number of participants with residual postinflammatory hyperpigmentation -burning sensation -wound dehiscence | 6 months
  redness or coloured pigmentation at wound site
Number of participants with burning sensation | 6 months
  feel burn at wound site
Number of participants with wound dehiscence(complete) | 6 months
  area of gaping of wound that requires secondary sutures
Number of participants with wound dehiscence(partial) | 6 months
  area of gaping of wound that requires frequent dressings only

CONTACTS AND LOCATIONS:
Overall Officials: Amira Dieb, MD, Principal Investigator — KasrAlainiH
Locations (1):
- KasralainiH, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No